CLINICAL TRIAL: NCT06999356
Title: Salud Diabetes: A Pilot Study Comparing Lifestyle Interventions and Real-Time Continuous Glucose Monitoring In Predominantly Hispanic/Latino Adults With Non-Insulin Treated Type 2 Diabetes And An HbA1c > 9%
Brief Title: Salud Diabetes: A Pilot Study Comparing Lifestyle Interventions and Real-Time Continuous Glucose Monitoring
Acronym: Salud Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sutter Health (Other)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024.099EXP; CMI-IIS-018 (Other Grant/Funding Number: Abbott)
Record Dates: First submitted 2025-05-12; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetes; Nutrition
Keywords: Type 2 Diabetes; Diabetes; Nutrition; Vegetables; Fruits
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fruits and Vegetables (Other): Fruits, Vegetables only and CGM devices
  Interventions: Device: CGM Device

INTERVENTIONS:
Device: CGM Device — Fruits and Vegetables and some groups will get CGM devices along with Fruits and Vegetables

SUMMARY:
The aim of this proposal is to determine the impact of a produce prescription program in predominantly Hispanic/Latino adults with established non-insulin treated T2D and an HbA1c at or above 9%.

DETAILED DESCRIPTION:
The aim of this proposal is to determine the impact of a produce prescription program in predominantly Hispanic/Latino adults with established non-insulin treated T2D and an HbA1c at or above 9%. For individuals not responding to the produce prescription program, they will be randomized to the addition of real-time continuous glucose monitoring (rtCGM) or continue with the produce prescription program only for a further 3 months.

ELIGIBILITY:
Inclusion Criteria: Adults (aged>18 years) with established T2D and HbA1c of 9% or higher per most recent test result within the last 6 months.

Agreement to only track glucose levels via study-provided CGM -

Exclusion Criteria: Type 1 diabetes, Insulin use, Pregnancy, Use of steroids or medications that impact glucose levels

Medications Include:

Atypical antipsychotics Clozapine Olanzapine Paliperidone Quietiapine Risperidone Corticosteroids Calcineurin inhibitors Cyclosporine Sirolimus Tacrolimus Protease Inhibitors Atazanavir Darunavir Fosamprenavir Indinavir Nelfinavir Ritonivir Saquinavir Tipranivir

Life expectancy less than 6 months Diagnosis of stage 5 kidney disease or at risk of needing dialysis per Investigator discretion Any active clinically significant disease or disorder which in the investigator's opinion could interfere with participation in the study.

Inability to follow study procedures per Investigator discretion

-

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c at 18 weeks compared to baseline | 18 weeks
  Change in HbA1c at 18 weeks compared to baseline

SECONDARY OUTCOMES:
Change in Body Weight | 6 weeks and 3 months
  Weight will be measured in kg.
Waist Circumference | 6 weeks and 3 months
  Waist Circumference will be measure in cm
Blood Pressure | 6 weeks and 3 months
  Blood pressure will be measure in mm Hg.
Depression and anxiety are measured using DASS-21 (Depression Anxiety Stress Scale - 21) | 6 weeks and 3 months
  For the scales, the DASS-21 (Depression Anxiety Stress Scale - 21) reports on depression, anxiety, and stress by using a self-report questionnaire with 21 items. It consists of three subscales, each with seven items, assessing the frequency and severity of symptoms related to each emotion.
  The questionnaire uses a Likert scale (0-3) where higher scores indicate greater symptom severity.
  Scoring: Each subscale (Depression, Anxiety, and Stress) is scored separately by summing the responses to its respective items. The total score for each subscale can range from 0 to 21.
  Interpretation: Higher scores on each subscale indicate a higher level of the corresponding variable.
Height | 6 weeks and 3 months.
  Height will be measure in inches.

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, PhD, Principal Investigator — Sutter Health
Locations (1):
- Sansum Clinic, Sutter Health, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Data set will be shared with the study team at Rice University for analysis of CGM data, demographics, and self-reported data. Direct identified will be removed but dates will be included
Supporting Information: ICF
Time Frame: May 2025
Access Criteria: Study team at Rice University

REFERENCES:
- [Background] Hernandez-Jimenez S, Garcia-Ulloa AC, Anaya P, Gasca-Pineda R, Sanchez-Trujillo LA, Pena Baca H, Gonzalez-Pier E, Graue-Hernandez EO, Aguilar-Salinas CA, Gomez-Perez FJ, Kershenobich-Stalnikowitz D; Group of Study CAIPaDi. Cost-effectiveness of a self-management and comprehensive training intervention in patients with type 2 diabetes up to 5 years of diagnosis in a specialized hospital in Mexico City. BMJ Open Diabetes Res Care. 2021 Jun;9(1):e002097. doi: 10.1136/bmjdrc-2020-002097. PMID 34167953
- [Background] Aiken M, Villa P, Lamotte M, Tewary V, Ramos M. Advancing glycemic management in people with diabetes; new approaches and measures. IQVIA Institute for Human Data Science Nov 2019. https://www.iqvia.com/insights/the-iqvia-institute/reports/advancing-glycemic-management-in-people-with-diabetes.
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Kerr D, Barua S, Glantz N, Conneely C, Kujan M, Bevier W, Larez A, Sabharwal A. Farming for life: impact of medical prescriptions for fresh vegetables on cardiometabolic health for adults with or at risk of type 2 diabetes in a predominantly Mexican-American population. BMJ Nutr Prev Health. 2020 Oct 5;3(2):239-246. doi: 10.1136/bmjnph-2020-000133. eCollection 2020 Dec. PMID 33521534
- [Background] Moon SJ, Kim KS, Lee WJ, Lee MY, Vigersky R, Park CY. Efficacy of intermittent short-term use of a real-time continuous glucose monitoring system in non-insulin-treated patients with type 2 diabetes: A randomized controlled trial. Diabetes Obes Metab. 2023 Jan;25(1):110-120. doi: 10.1111/dom.14852. Epub 2022 Sep 23. PMID 36053813
- [Background] Wada E, Onoue T, Kobayashi T, Handa T, Hayase A, Ito M, Furukawa M, Okuji T, Okada N, Iwama S, Sugiyama M, Tsunekawa T, Takagi H, Hagiwara D, Ito Y, Suga H, Banno R, Kuwatsuka Y, Ando M, Goto M, Arima H. Flash glucose monitoring helps achieve better glycemic control than conventional self-monitoring of blood glucose in non-insulin-treated type 2 diabetes: a randomized controlled trial. BMJ Open Diabetes Res Care. 2020 Jun;8(1):e001115. doi: 10.1136/bmjdrc-2019-001115. PMID 32518063
- [Background] Vigersky RA, Fonda SJ, Chellappa M, Walker MS, Ehrhardt NM. Short- and long-term effects of real-time continuous glucose monitoring in patients with type 2 diabetes. Diabetes Care. 2012 Jan;35(1):32-8. doi: 10.2337/dc11-1438. Epub 2011 Nov 18. PMID 22100963
- [Background] Glantz NM, Duncan I, Ahmed T, Fan L, Reed BL, Kalirai S, Kerr D. Racial and Ethnic Disparities in the Burden and Cost of Diabetes for US Medicare Beneficiaries. Health Equity. 2019 May 15;3(1):211-218. doi: 10.1089/heq.2019.0004. eCollection 2019. PMID 31289781
- [Background] Davies MJ, Aroda VR, Collins BS, Gabbay RA, Green J, Maruthur NM, Rosas SE, Del Prato S, Mathieu C, Mingrone G, Rossing P, Tankova T, Tsapas A, Buse JB. Management of Hyperglycemia in Type 2 Diabetes, 2022. A Consensus Report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2022 Nov 1;45(11):2753-2786. doi: 10.2337/dci22-0034. PMID 36148880
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S140-S157. doi: 10.2337/dc23-S009. PMID 36507650
- [Background] Pednekar P, Heller DA, Peterson AM. Association of Medication Adherence with Hospital Utilization and Costs Among Elderly with Diabetes Enrolled in a State Pharmaceutical Assistance Program. J Manag Care Spec Pharm. 2020 Sep;26(9):1099-1108. doi: 10.18553/jmcp.2020.26.9.1099. PMID 32857648
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Background] Centers for Disease Control and Prevention. National Diabetes Statistics Report: Estimates of Diabetes and Its Burden in the United States, 2014 (1st ed.). 2014. Atlanta, GA: Department of Health and Human Services; Available at https://cdc.gov/diabetes/pubs/statsreport14/national-diabetes-report-web.pdf